CLINICAL TRIAL: NCT07337707
Title: New Microbiota-endocrine Axis in Fructose Malabsorption-caused Visceral Hypersensitivity in Irritable Bowel Syndrome.
Acronym: ENDOLORII
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Collaborators: ANR AAPG2023 (Unknown); INRAE-Micalis AMIPEM (Unknown); INRAE-Micalis FINE (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023/0252/HP
Record Dates: First submitted 2025-07-02; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Irritable Bowel Syndrome (IBS)
Keywords: visceral hypersensitivity; fructose malabsorption; microbiota
MeSH Terms: conditions — Irritable Bowel Syndrome; Fructose Intolerance | interventions — Lactulose; Hematologic Tests; Diet Records

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- MalF-HyperSens (Experimental): Patients with IBS with fructose malabsorption and with visceral hypersensitivity
  Interventions: Biological: urine intestinal permeability test or lactulose/mannitol test; Biological: Blood test; Other: food diary; Other: stool samples; Other: Microbiota analysis
- MalF-NormoSens (Experimental): Patients with IBS with fructose malabsorption and without hypersensitivity
  Interventions: Biological: urine intestinal permeability test or lactulose/mannitol test; Biological: Blood test; Other: food diary; Other: stool samples; Other: Microbiota analysis
- NormoF-HyperSens (Experimental): Patients with IBS without fructose malabsorption and with visceral hypersensitivity
  Interventions: Biological: urine intestinal permeability test or lactulose/mannitol test; Biological: Blood test; Other: food diary; Other: stool samples; Other: Microbiota analysis
- NormoF-NormoSens (Experimental): Patients with IBS without fructose malabsorption and without visceral hypersensitivity
  Interventions: Biological: urine intestinal permeability test or lactulose/mannitol test; Biological: Blood test; Other: food diary; Other: stool samples; Other: Microbiota analysis

INTERVENTIONS:
Biological: urine intestinal permeability test or lactulose/mannitol test — Patients will be required to fast for 12 hours and, after emptying their bladder, patients will be asked to drink 100 mL of water containing 10 g of lactulose and 5 g of mannitol. At the patient's inclusion visit, and before the test at the V1 follow-up visit, the patient will be given an explanation with recommendations on their food intake in the 24 hours before and 24 hours during the test (urine collection). Patients will be asked not to drink for 2 hours and not to eat for 5 hours after taking the lactulose and mannitol. An exhaustive urine collection will then be carried out at the patient's home over the 24 hours following the intake of the sugars. The 24-hour urine will be collected in a plastic 24-hour urine container suitable for hospital use. This urine collection will be brought back for visit 2 the following day. On receipt of the urine, the volume of urine will be noted and the appearance of the urine recorded and stored before analysis.
Biological: Blood test — A fasting blood sample will be taken in 1 x 4ml EDTA-Aprotinin tube on the morning of the urine test (V1 follow-up visit). The tube will be centrifuged within 15 minutes at 4°C and then aliquoted into 3 x 500μL tubes which will be immediately frozen at -80°C for storage in a biocollection with a view to later measuring gastrointestinal peptides such as CCK, neurotensin and GLP-1.
Other: food diary — On the day of inclusion, all patients were given a food diary to fill in. They will have to fill it in over a period of 4 days, including 1 weekend day. They will be asked to note down all the food they eat during this period, as well as the quantities. The diary will be collected at the V1 visit and will then be analysed by a dietician, who will assess the average daily consumption of fructose in g/d (total fructose consumption, consumption of fructose in excess of glucose, dietary origin of fructose).
Other: stool samples — All patients will have their stools collected. Patients will have their stool collected at home using a collector given to them at the inclusion visit. They will have to bring back the stool within 6 hours for preparation and storage at -80°C.
Other: Microbiota analysis — Stools will be used to analyse the composition of the intestinal microbiota by sequencing amplicons from the V3-V4 region of bacterial 16S rRNA.

SUMMARY:
Irritable bowel syndrome (IBS) affects around 4% of the general population and remains the most common functional bowel disorder. It is defined by the Rome criteria as the presence of abdominal pain associated with transit disorders. The impact on quality of life and the associated costs make it a public health problem.

Visceral hypersensitivity is one of the functional markers of the disease and plays a part in the genesis of symptoms. It could therefore also be a therapeutic target to be explored. Diet and the intestinal microbiota are also part of the recognised pathophysiological mechanisms of this disease. Carbohydrates malabsorbed by the intestine are metabolised by the microbiota, which may contribute to the genesis of symptoms. Among these carbohydrates, fructose appears to be of particular interest. Its absorption capacity is limited, yet fructose consumption is increasing. Fructose malabsorption at a dose of 25 g is present in 22% of IBS patients. Fructose malabsorption is also associated with visceral hypersensitivity. However, the mechanism of this association remains unknown. In models of malabsorbed mice with visceral hypersensitivity, an increase in cholecystokinin was found in the terminal ileum and cecum, suggesting a potential role for this hormone in this model of IBS. However, the underlying mechanism remains poorly understood.

The objective is to determine if microbiota signature is specific of visceral hypersensitivity associated with fructose malabsorption in IBS patients.

60 patients with IBS will be included in the study in 4 groups:

1. n=15 patients with visceral hypersensitivity and fructose malabsorption
2. n=15 patients with visceral hypersensitivity and without fructose malabsorption
3. n=15 patients without visceral hypersensitivity and with fructose malabsorption
4. n=15 patients without visceral hypersensitivity and without fructose malabsorption

All patients will filled validated questionnaires and 4-days food diary. They will also have a urinary permeability test (lactulose/mannitol test) and collected stools samples for microbiota analysis.

ELIGIBILITY:
Inclusion Criteria:

For all groups:

* Patients with IBS defined by current Rome criteria (currently IV)
* Adult, aged 18 to 75
* Regulatory criteria :

  * Membership of a social security scheme
  * Adult having read and understood the information letter and signed the consent form
  * Woman of childbearing age with effective contraception for the duration of the study such as oestroprogestins, intrauterine device, tubal ligation, vasectomised partner or sexual abstinence (no heterosexual intercourse for 1 month and a negative urine pregnancy test at inclusion).
  * Postmenopausal women: confirmatory diagnosis (non-medically induced amenorrhoea for at least 12 months prior to the inclusion visit or biologically documented)
  * Women of childbearing age who have been rendered surgically infertile (e.g. hysterectomy, bilateral salpingectomy, bilateral oophorectomy).

For the IBS group with fructose malabsorption and visceral hypersensitivity (named group of interest, MalF-HyperSens) (1):

* 25g fructose breath test in favour of fructose malabsorption
* Rectal barostat finding visceral hypersensitivity

For the IBS group with fructose malabsorption and without visceral hypersensitivity (known as the MalF-NormoSens group) (2):

* Fructose breath test at 25g dose in favour of fructose malabsorption
* Rectal barostat finding no visceral hypersensitivity

For the IBS group without fructose malabsorption and visceral hypersensitivity (named NormoF-HyperSens group) (3):

* Fructose breath test at 25g dose in favour of no fructose malabsorption
* Rectal barostat finding visceral hypersensitivity

For the IBS group without fructose malabsorption or visceral hypersensitivity (called the NormoF-NormoSens group) (4):

* Fructose breath test at a dose of 25g in favour of the absence of fructose malabsorption
* Rectal barostat finding no visceral hypersensitivity

Exclusion Criteria:

* Patient who has not undergone a fructose breath test or a barostat in our department in the last 10 years.
* Patient with organic digestive pathology (chronic inflammatory bowel disease, microscopic colitis, digestive cancer, celiac disease)
* Systemic antibiotic use (oral, IV or IM) in the month prior to inclusion
* Regulatory criteria :

  * Pregnant or parturient or breast-feeding woman or proven absence of contraception,
  * Person deprived of liberty by an administrative or judicial decision or person placed under court protection / sub- guardianship or curatorship,
  * Person undergoing research participating in another trial / having participated in another trial within a period of 2 weeks,
  * History of illness or psychological or sensory abnormality likely to prevent the subject from fully understanding the conditions required for participation in the protocol or preventing him/her from giving informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
microbiota analysis | from enrollment up to 18 months
  16S RNA gene sequencing
metabolites analysis | from enrollment up to 18 months
  Mass spectrometry-based metabolomics

SECONDARY OUTCOMES:
Intestinal permeability | from enrollment up to 18 months
  lactulose-mannitol test
low grade inflammation | from enrollment up to 18 months
  fecal calprotectin
fructose consumption | from enrollment up to 18 months
  delay fructose consumption (g/D)
IBS severity | from enrollment up to 18 months
  IBS-SSS
Stool consistency | from enrollment up to 18 months
  Bristol stool form
anxiety | from enrollment up to 18 months
  STAI
psychological distress | from enrollment up to 18 months
  HAD
impact on quality of life | from enrollment up to 18 months
  IBSQOL

CONTACTS AND LOCATIONS:
Overall Officials: MELCHIOR Pr MELCHIOR, Principal Investigator — University Hospital, Rouen
Locations (1):
- CHU de Rouen, Rouen, France

IPD SHARING:
Plan to Share IPD: No